CLINICAL TRIAL: NCT00392639
Title: Clinical Interest of Endovascular Cooling in the Management of Cardiac Arrest: Impact on Mortality in a Randomized Medico-economical Trial (the ICEREA Study)
Brief Title: Clinical and Economical Interest of Endovascular Cooling in the Management of Cardiac Arrest (ICEREA Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Alsius Corporation (Industry); distributed in France by (Ambiguous); IST Cardiology (Le Fresne Camilly, France) (Unknown)
Responsible Party: Mathieu QUINTIN, Department Clinical Research of Developpement
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P051038
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2007-07

CONDITIONS: Hypothermia; Heart Arrest
Keywords: Heart arrest; Cardiopulmonary resuscitation; Humans; Hypothermia; Brain diseases; Hypoxia-ischemia; Cost Benefit Analysis; Prospective study; Comparative study; Treatment outcome; Hypothermia for; out-of-hospital cardiac arrest; from cardiac origin; successfully resuscitated
MeSH Terms: conditions — Hypothermia; Heart Arrest; Brain Diseases; Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1-2 (Experimental): Comparison of 2 cooling procedures
  Interventions: Procedure: Comparison of 2 cooling procedures

INTERVENTIONS:
Procedure: Comparison of 2 cooling procedures — Comparison of 2 cooling procedures

SUMMARY:
According to international guidelines, mild therapeutic hypothermia is recommended for resuscitated patients after cardiac arrest due to ventricular fibrillation. Whether external or internal cooling is superior in terms of prognosis or security remains unknown. The aim of this study is to evaluate in a randomized trial the clinical and economical interests of the endovascular cooling versus the conventional external cooling for the management of hypothermia after cardiac arrest.

DETAILED DESCRIPTION:
According to international guidelines, mild therapeutic hypothermia is recommended for resuscitated patients after experiencing cardiac arrest from cardiac origin: "unconscious adult patients with spontaneous circulation after cardiac arrest should be cooled to 32-34°C for 12-24 hours when the initial rhythm was ventricular fibrillation" or pulseless ventricular tachycardia. "Such cooling may also be beneficial for other rhythm or in-hospital cardiac arrest".

"External or internal cooling techniques can be used to initiate cooling within minutes to hours". The two main randomized and positive studies dealing with the efficiency of hypothermia after cardiac arrest have used external cooling systems. However, several animal studies documented the importance of initiating hypothermia as soon as possible after cardiac arrest. Intravascular cooling enables more rapid induction of hypothermia compared with external cooling method after brain injury. Although several human studies have also documented that intravascular cooling provides more precise control of core temperature than external methods and although an endovascular method has been used safely in pilot studies in those experiencing hypothermia after cardiac arrest, the superiority of such a cooling on the prognosis after cardiac arrest remains unknown, as well as its cost efficiency.

The aim of this study is to evaluate in a randomized trial the potential clinical and economical interests of the endovascular cooling versus the conventional external cooling for the management of cardiac arrest from cardiac origin. With a clinical primary endpoint (survival without major neurological sequels), this study will also focus on important secondary endpoints, as the burden of nurse work and the economical costs induced by these 2 different methods of cooling.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 79 years old
* Out-of-hospital cardiac arrest (OH-CA) due to a presumed cardiac etiology
* Delay between OH-CA and return of spontaneous circulation (ROSC) < 60 minutes
* Delay between ROSC and starting cooling < 240 minutes
* Patient not obeying verbal command after ROSC and prior to starting cooling
* Availability of the "CoolGard" device (ALSIUS product)

Exclusion Criteria:

* Do not reanimate order or terminal disease before inclusion
* Known pregnancy
* Clinical hemorrhagic syndrome or known coagulopathy
* Contra-indication to device usage (such as femoral venous access impossible)
* Hypothermia at admission < 30°C
* Etiology of OH-CA thought to be extra-cardiac (trauma, bleeding or anoxia)
* In hospital cardiac arrest
* Refractory shock (need for extra-corporeal life support)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2006-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Clinical interest of endovascular cooling versus conventional external cooling for the management of cardiac arrest from cardiac origin | 28 days

SECONDARY OUTCOMES:
Cost/efficiency ratio (endovascular versus conventional cooling) | at 28 days
Evaluation of the paramedical burden of work | at 28 days
Evaluation of the nurse's satisfaction index | at 28 days
Evaluation of treatment costs: global costs and costs within the first 48 hours of hospitalization | at 28 days
Time necessary to reach the target temperature (33°C): mean speed of temperature decrease | at 28 days
deviations of more than 1°C compared with the target temperature during the 24 hours (24H) after reaching that target temperature | at 28 days
mean speed of rewarming | at 28 days
Safety of the method (type of adverse events) | at 28 days
Analysis according to the type and the cause of the cardiac arrest, duration of resuscitation maneuvers, success of coronary angioplasty, number of organ failures (Logistic Organ Dysfunction System [LODS] | at 28 days
Sequential Organ Failure Assessment [SOFA] | at 28 days
and Organ Dysfunctions and/or Infection [ODIN] scores | at 28 days
Simplified Acute Physiology [SAPS II]), duration of Intensive Care Unit (ICU) stay and duration of mechanical ventilation | at 28 days
The efficiency is measured on survival and on better neurological outcome, as defined by CPC 1 or 2 on the Pittsburgh cerebral performance categories (CPC), with an expected 12% improvement of the survival without major sequels at day 28 after inclusion. | at 28 days and 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Frederic BAUD, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Teaching Lariboisière Hospital, Paris, France

REFERENCES:
- [Result] Bernard SA, Gray TW, Buist MD, Jones BM, Silvester W, Gutteridge G, Smith K. Treatment of comatose survivors of out-of-hospital cardiac arrest with induced hypothermia. N Engl J Med. 2002 Feb 21;346(8):557-63. doi: 10.1056/NEJMoa003289. PMID 11856794
- [Result] Hypothermia after Cardiac Arrest Study Group. Mild therapeutic hypothermia to improve the neurologic outcome after cardiac arrest. N Engl J Med. 2002 Feb 21;346(8):549-56. doi: 10.1056/NEJMoa012689. PMID 11856793
- [Result] Nolan JP, Morley PT, Vanden Hoek TL, Hickey RW, Kloeck WG, Billi J, Bottiger BW, Morley PT, Nolan JP, Okada K, Reyes C, Shuster M, Steen PA, Weil MH, Wenzel V, Hickey RW, Carli P, Vanden Hoek TL, Atkins D; International Liaison Committee on Resuscitation. Therapeutic hypothermia after cardiac arrest: an advisory statement by the advanced life support task force of the International Liaison Committee on Resuscitation. Circulation. 2003 Jul 8;108(1):118-21. doi: 10.1161/01.CIR.0000079019.02601.90. No abstract available. PMID 12847056
- [Result] International Liaison Committee on Resuscitation. 2005 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science with Treatment Recommendations. Part 4: Advanced life support. Resuscitation. 2005 Nov-Dec;67(2-3):213-47. doi: 10.1016/j.resuscitation.2005.09.018. No abstract available. PMID 16324990
- [Result] Steinberg GK, Ogilvy CS, Shuer LM, Connolly ES Jr, Solomon RA, Lam A, Kassell NF, Baker CJ, Giannotta SL, Cockroft KM, Bell-Stephens TE, Allgren RL. Comparison of endovascular and surface cooling during unruptured cerebral aneurysm repair. Neurosurgery. 2004 Aug;55(2):307-14; discussion 314-5. doi: 10.1227/01.neu.0000129683.99430.8c. PMID 15271236
- [Result] Al-Senani FM, Graffagnino C, Grotta JC, Saiki R, Wood D, Chung W, Palmer G, Collins KA. A prospective, multicenter pilot study to evaluate the feasibility and safety of using the CoolGard System and Icy catheter following cardiac arrest. Resuscitation. 2004 Aug;62(2):143-50. doi: 10.1016/j.resuscitation.2004.02.016. PMID 15294399
- [Derived] Deye N, Cariou A, Girardie P, Pichon N, Megarbane B, Midez P, Tonnelier JM, Boulain T, Outin H, Delahaye A, Cravoisy A, Mercat A, Blanc P, Santre C, Quintard H, Brivet F, Charpentier J, Garrigue D, Francois B, Quenot JP, Vincent F, Gueugniaud PY, Mira JP, Carli P, Vicaut E, Baud FJ; Clinical and Economical Impact of Endovascular Cooling in the Management of Cardiac Arrest (ICEREA) Study Group. Endovascular Versus External Targeted Temperature Management for Patients With Out-of-Hospital Cardiac Arrest: A Randomized, Controlled Study. Circulation. 2015 Jul 21;132(3):182-93. doi: 10.1161/CIRCULATIONAHA.114.012805. Epub 2015 Jun 19. PMID 26092673